CLINICAL TRIAL: NCT01829295
Title: First-line Antimetabolites as Steroid-sparing Treatment (FAST) Uveitis Trial
Brief Title: Methotrexate and Mycophenolate Mofetil for UVEITIS
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other); Oregon Health and Science University (Other); Asociación para Evitar la Ceguera en México (Other); Royal Victoria Eye and Ear Hospital (Other Government); Northwestern University (Other); National Eye Institute (NEI) (NIH); King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-08227; 5U10EY021125 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Uveitis
Keywords: antimetabolite, noninfectious
MeSH Terms: conditions — Uveitis | interventions — Mycophenolic Acid; Methotrexate; Prednisone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): oral methotrexate
  Interventions: Drug: Methotrexate; Drug: Prednisone
- Mycophenolate Mofetil (Experimental): oral mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate mofetil — For the first two weeks, an introductory dose of 500 mg twice a day (BID) orally. After two weeks, the dose will be increased to 1.5 g BID.
  Other Names: Cellcept
  Arms: Mycophenolate Mofetil
Drug: Methotrexate — For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Arms: Methotrexate
Drug: Prednisone — All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.

SUMMARY:
In the First-line Antimetabolites as Steroid-sparing Treatment (FAST) Uveitis Trial, the investigators propose to establish which immunosuppressive therapy, methotrexate or mycophenolate mofetil, is more effective as a first-line, corticosteroid-sparing agent for the treatment of non-infectious uveitis in a block-randomized, observer-masked, comparative effectiveness trial.

DETAILED DESCRIPTION:
This is a randomized comparative effectiveness trial to determine which treatment, methotrexate or mycophenolate mofetil, is more effective as first-line corticosteroid-sparing treatment for patients with non-infectious intermediate, posterior and panuveitis requiring corticosteroid-sparing therapy. The primary outcome is treatment success assessed at the 6 month visit (Phase 1, 0-6 months). If patients are a treatment success, they continue on the medication for another 6 months (Phase 1, 6-12 months). Patients who are a treatment failure can crossover to the other medication (Phase 2, 0-6 months).

ELIGIBILITY:
Inclusion Criteria:

* All the following criteria must be met at enrollment:

Historical non-infectious intermediate, anterior and intermediate, posterior or panuveitis in at least one eye

Active inflammation within the last 180 days, defined by the presence of any of the following (in at least one eye) according to Standardization of Uveitis Nomenclature (SUN) criteria:

* ≥ 2+ anterior chamber cells
* ≥ 2+ vitreous haze
* active retinal or choroidal lesions

Active inflammation at enrollment, defined by the presence of any of the following (in at least one eye) according to SUN criteria:

* ≥1+ anterior chamber cells and/or
* ≥1+ vitreous haze and/or
* active retinal/choroidal lesions

At least one of the following criteria must be met before or at enrollment:

* Active inflammation after 4 weeks of high-dose (1mg/kg prednisone equivalent) corticosteroid treatment or 4 weeks following a regional corticosteroid injection
* Treatment with oral corticosteroids resulting in a reduction of inflammation, followed by an increase in inflammation (of at least 1 grade in anterior chamber cells or vitreous haze or a change of non-active to active lesions) when corticosteroid is tapered, in the 180 weeks prior to enrollment
* Active inflammation after long-acting corticosteroid injection 4 weeks to 180 days prior to enrollment
* Active inflammation after treatment with >10mg/day oral prednisone for at least the past 90 days prior to enrollment
* Known chronic condition necessitating corticosteroid-sparing immunosuppressive treatment: Behcet's disease with posterior segment involvement, multifocal choroiditis with panuveitis, serpiginous choroidopathy, birdshot retinochoroidopathy, diffuse retinal vasculitis, Vogt-Koyanagi-Harada with bullous serous retinal detachments and/or choroidal detachments, sympathetic ophthalmia. No prior therapy required for these patients

Willingness to start corticosteroid treatment at 1mg/kg or 60mg a day of prednisone, whichever is less

Willingness to limit alcohol consumption

Willingness to use an acceptable method of contraception during the study period (i.e. pharmacologic medications, devices, barrier methods) or abstinence.

* Exclusion Criteria: Any of the following

Any infectious cause of uveitis

Prior immunosuppressive therapy other than corticosteroids in the past 12 months

Prior intolerability or safety issues with methotrexate or mycophenolate mofetil

Prior failure to control ocular or other inflammation using methotrexate or mycophenolate mofetil

Prior biologic therapy at any time

Media opacity (such as cataract and/or corneal scar) and/or extensive posterior synechiae such that examination of the posterior segment is not possible in both eyes

Chronic hypotony (IOP < 5 mm Hg for > 3 months) in both eyes

Periocular or intravitreal corticosteroid injection in the past 4 weeks

Fluocinolone acetonide implant in either eye in < 3 years

Intraocular surgery in < 30 days, or planning on getting surgery within the next 6 months

Best spectacle-corrected visual acuity (BSCVA) of hand motions or worse in better eye

< 16 years of age at enrollment

Planning to conceive during the study period, pregnant or breast-feeding (blood or urine pregnancy test for all females, excluding those who are post-menopausal is mandatory)*

Any history of cancer (If a patient has a history of non-melanoma skin cancer they can still be considered for inclusion in this study, provided it is not currently active).

Systemic autoimmune disease anticipated to dictate treatment course

Abnormal Complete blood count (≤ 2,500 white blood cells and/or ≤ 75,000 platelets and/or ≤9 hemoglobin) within 4 weeks prior to enrollment*

Abnormal alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal for the lab and/or creatinine ≥ 1.5 within 4 weeks prior to enrollment*

Evidence of active tuberculosis, HIV infection, syphilis, or hepatitis B or C (patients must have a tuberculin skin test, or interferon-gamma release assay, a chest radiograph, Rapid plasma reagin / Venereal disease research laboratory test (RPR/VDRL), fluorescent treponemal antibody absorption test (FTA-ABS), or other treponemal tests, Hepatitis B surface antigen, Hepatitis C antibody tests, and HIV test within 90 days prior to enrollment)**

*Testing required within 4 weeks prior to enrollment; **Testing required within 90 days prior to enrollment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-08; Primary Completion 2018-02-21 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Acharya, MD, MS, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (3):
  - Francis I Proctor Foundation, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Oregon Health and Science University - Casey Eye Institute, Portland, Oregon
- Royal Victorian Eye and Ear Hospital, Melbourne, Victoria, Australia
- India (3):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu
- Asociacion Para Evita La Ceguera en Mexico, Mexico City, Mexico City, Mexico
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Galor A, Jabs DA, Leder HA, Kedhar SR, Dunn JP, Peters GB 3rd, Thorne JE. Comparison of antimetabolite drugs as corticosteroid-sparing therapy for noninfectious ocular inflammation. Ophthalmology. 2008 Oct;115(10):1826-32. doi: 10.1016/j.ophtha.2008.04.026. Epub 2008 Jun 25. PMID 18579209
- [Background] Siepmann K, Huber M, Stubiger N, Deuter C, Zierhut M. Mycophenolate mofetil is a highly effective and safe immunosuppressive agent for the treatment of uveitis : a retrospective analysis of 106 patients. Graefes Arch Clin Exp Ophthalmol. 2006 Jul;244(7):788-94. doi: 10.1007/s00417-005-0066-8. Epub 2005 Sep 15. PMID 16163494
- [Background] Teoh SC, Hogan AC, Dick AD, Lee RW. Mycophenolate mofetil for the treatment of uveitis. Am J Ophthalmol. 2008 Nov;146(5):752-60, 760.e1-3. doi: 10.1016/j.ajo.2008.03.004. Epub 2008 May 2. PMID 18455143
- [Background] Thorne JE, Jabs DA, Qazi FA, Nguyen QD, Kempen JH, Dunn JP. Mycophenolate mofetil therapy for inflammatory eye disease. Ophthalmology. 2005 Aug;112(8):1472-7. doi: 10.1016/j.ophtha.2005.02.020. PMID 16061096
- [Background] Larkin G, Lightman S. Mycophenolate mofetil. A useful immunosuppressive in inflammatory eye disease. Ophthalmology. 1999 Feb;106(2):370-4. doi: 10.1016/S0161-6420(99)90078-7. PMID 9951492
- [Background] Baltatzis S, Tufail F, Yu EN, Vredeveld CM, Foster CS. Mycophenolate mofetil as an immunomodulatory agent in the treatment of chronic ocular inflammatory disorders. Ophthalmology. 2003 May;110(5):1061-5. doi: 10.1016/S0161-6420(03)00092-7. PMID 12750115
- [Background] Choudhary A, Harding SP, Bucknall RC, Pearce IA. Mycophenolate mofetil as an immunosuppressive agent in refractory inflammatory eye disease. J Ocul Pharmacol Ther. 2006 Jun;22(3):168-75. doi: 10.1089/jop.2006.22.168. PMID 16808677
- [Background] Bom S, Zamiri P, Lightman S. Use of methotrexate in the management of sight-threatening uveitis. Ocul Immunol Inflamm. 2001 Mar;9(1):35-40. doi: 10.1076/ocii.9.1.35.3983. PMID 11262666
- [Background] Dev S, McCallum RM, Jaffe GJ. Methotrexate treatment for sarcoid-associated panuveitis. Ophthalmology. 1999 Jan;106(1):111-8. doi: 10.1016/S0161-6420(99)90011-8. PMID 9917790
- [Background] Foeldvari I, Wierk A. Methotrexate is an effective treatment for chronic uveitis associated with juvenile idiopathic arthritis. J Rheumatol. 2005 Feb;32(2):362-5. PMID 15693100
- [Background] Gangaputra S, Newcomb CW, Liesegang TL, Kacmaz RO, Jabs DA, Levy-Clarke GA, Nussenblatt RB, Rosenbaum JT, Suhler EB, Thorne JE, Foster CS, Kempen JH; Systemic Immunosuppressive Therapy for Eye Diseases Cohort Study. Methotrexate for ocular inflammatory diseases. Ophthalmology. 2009 Nov;116(11):2188-98.e1. doi: 10.1016/j.ophtha.2009.04.020. Epub 2009 Sep 12. PMID 19748676
- [Background] Holz FG, Krastel H, Breitbart A, Schwarz-Eywill M, Pezzutto A, Volcker HE. Low-dose methotrexate treatment in noninfectious uveitis resistant to corticosteroids. Ger J Ophthalmol. 1992;1(3-4):142-4. PMID 1483126
- [Background] Shah SS, Lowder CY, Schmitt MA, Wilke WS, Kosmorsky GS, Meisler DM. Low-dose methotrexate therapy for ocular inflammatory disease. Ophthalmology. 1992 Sep;99(9):1419-23. doi: 10.1016/s0161-6420(92)31790-7. PMID 1407973
- [Background] Taylor SR, Habot-Wilner Z, Pacheco P, Lightman SL. Intraocular methotrexate in the treatment of uveitis and uveitic cystoid macular edema. Ophthalmology. 2009 Apr;116(4):797-801. doi: 10.1016/j.ophtha.2008.10.033. PMID 19344827
- [Background] Daniel E, Thorne JE, Newcomb CW, Pujari SS, Kacmaz RO, Levy-Clarke GA, Nussenblatt RB, Rosenbaum JT, Suhler EB, Foster CS, Jabs DA, Kempen JH. Mycophenolate mofetil for ocular inflammation. Am J Ophthalmol. 2010 Mar;149(3):423-32.e1-2. doi: 10.1016/j.ajo.2009.09.026. Epub 2009 Dec 30. PMID 20042178
- [Background] Sobrin L, Christen W, Foster CS. Mycophenolate mofetil after methotrexate failure or intolerance in the treatment of scleritis and uveitis. Ophthalmology. 2008 Aug;115(8):1416-21, 1421.e1. doi: 10.1016/j.ophtha.2007.12.011. Epub 2008 Jan 25. PMID 18221998
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Jabs DA, Rosenbaum JT, Foster CS, Holland GN, Jaffe GJ, Louie JS, Nussenblatt RB, Stiehm ER, Tessler H, Van Gelder RN, Whitcup SM, Yocum D. Guidelines for the use of immunosuppressive drugs in patients with ocular inflammatory disorders: recommendations of an expert panel. Am J Ophthalmol. 2000 Oct;130(4):492-513. doi: 10.1016/s0002-9394(00)00659-0. PMID 11024423
- [Result] Reddy AK, Miller DC, Sura AA, Rathinam SR, Gonzales JA, Thundikandy R, Kanakath A, Murugan B, Vedhanayaki R, Lim LL, Suhler EB, Doan T, Al-Dhibi HA, Goldstein DA, Arellanes-Garcia L, Acharya NR. Risk of failing both methotrexate and mycophenolate mofetil from the First-line Antimetabolites as Steroid-sparing Treatment (FAST) uveitis trial. J Ophthalmic Inflamm Infect. 2023 Jun 9;13(1):29. doi: 10.1186/s12348-023-00350-5. PMID 37294447
- [Result] Chattopadhyay A, Rathinam SR, Gonzales JA, Kelly NK, Thundikandy R, Kanakath A, Murugan SB, Vedhanayaki R, Lim LL, Suhler EB, Al-Dhibi HA, Doan T, Ebert CD, Porco TC, Acharya NR; FAST Research Group. Association between Quality of Life and Visual Acuity in a Randomized Clinical Trial of Patients with Uveitis Taking Antimetabolites. Ocul Immunol Inflamm. 2024 Apr;32(3):301-309. doi: 10.1080/09273948.2023.2169714. Epub 2023 Feb 7. PMID 36749914
- [Result] Sura AA, Sun Y, Reddy AK, Rathinam SR, Gonzales JA, Thundikandy R, Vedhanayaki R, Kanakath A, Murugan B, Doan TA, Lim LL, Suhler EB, Al-Dhibi HA, Acharya NR; FAST Research Group. Reduced Dose Methotrexate and Mycophenolate Mofetil in Noninfectious Uveitis: A Sub-Analysis from the First-Line Antimetabolites as Steroid Sparing Therapy (FAST) Trial. Ocul Immunol Inflamm. 2024 Aug;32(6):955-960. doi: 10.1080/09273948.2023.2165949. Epub 2023 Jan 26. PMID 36701644
- [Result] Tsui E, Rathinam SR, Gonzales JA, Thundikandy R, Kanakath A, Balamurugan S, Vedhanayaki R, Lim LL, Suhler EB, Al-Dhibi HA, Doan T, Keenan J, Ebert CD, Kim E, Madow B, Porco TC, Acharya NR; FAST Research Group. Outcomes of Uveitic Macular Edema in the First-line Antimetabolites as Steroid-Sparing Treatment Uveitis Trial. Ophthalmology. 2022 Jun;129(6):661-667. doi: 10.1016/j.ophtha.2022.02.002. Epub 2022 Feb 8. PMID 35143800
- [Result] Kelly NK, Chattopadhyay A, Rathinam SR, Gonzales JA, Thundikandy R, Kanakath A, Murugan SB, Vedhanayaki R, Cugley D, Lim LL, Suhler EB, Al-Dhibi HA, Ebert CD, Berlinberg EJ, Porco TC, Acharya NR; FAST Research Group. Health- and Vision-Related Quality of Life in a Randomized Controlled Trial Comparing Methotrexate and Mycophenolate Mofetil for Uveitis. Ophthalmology. 2021 Sep;128(9):1337-1345. doi: 10.1016/j.ophtha.2021.02.024. Epub 2021 Mar 4. PMID 33675850
- [Result] Kong CL, Kelly NK, Sundararajan M, Rathinam SR, Gonzales JA, Thundikandy R, Vedhanayaki R, Kanakath A, Murugan B, Doan T, Goldstein D, Al-Dhibi HA, Acharya NR. Comparison of CD4 Counts with Mycophenolate Mofetil versus Methotrexate from the First-line Antimetabolites as Steroid-sparing Treatment (FAST) Uveitis Trial. Ocul Immunol Inflamm. 2022 Jan 2;30(1):198-202. doi: 10.1080/09273948.2020.1774906. Epub 2020 Aug 11. PMID 32779952
- [Result] Rathinam SR, Gonzales JA, Thundikandy R, Kanakath A, Murugan SB, Vedhanayaki R, Lim LL, Suhler EB, Al-Dhibi HA, Doan T, Keenan JD, Rao MM, Ebert CD, Nguyen HH, Kim E, Porco TC, Acharya NR; FAST Research Group. Effect of Corticosteroid-Sparing Treatment With Mycophenolate Mofetil vs Methotrexate on Inflammation in Patients With Uveitis: A Randomized Clinical Trial. JAMA. 2019 Sep 10;322(10):936-945. doi: 10.1001/jama.2019.12618. PMID 31503307
- [Result] Bui AD, Kong CL, Kelly NK, Rathinam SR, Gonzales JA, Thundikandy R, Kanakath A, Murugan B, Vedhanayaki R, Lim LL, Suhler EB, Al-Dhibi HA, Doan T, Acharya NR; First-Line Antimetabolites as Steroid-Sparing Treatment Research Group. Time to Uveitis Control with Methotrexate and Mycophenolate Mofetil. Ophthalmology. 2022 Jun;129(6):721-723. doi: 10.1016/j.ophtha.2022.01.020. Epub 2022 Jan 25. No abstract available. PMID 35085661
- [Derived] Sundararajan M, Rathinam SR, Thundikandy R, Kanakath A, Balamurugan S, Vedhanayaki R, Miller DC, Lim LL, Suhler EB, Al-Dhibi HA, Arellanes-Garcia L, Reddy AK, Feng S, Doan T, Porco TC, Shantha JG, Acharya NR, Gonzales JA. Association Between Baseline Macular Morphologic Features on Optical Coherence Tomography and Visual Outcomes in Patients with Vogt-Koyanagi-Harada Disease. Ocul Immunol Inflamm. 2025 Feb;33(2):263-270. doi: 10.1080/09273948.2024.2391420. Epub 2024 Aug 27. PMID 39190826

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate Only: oral methotrexate
  Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg twice a day (BID) once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
  These patients never switched over to receive mycophenolate mofetil as they were a treatment success at Month 6.
- Mycophenolate Mofetil Only: oral mycophenolate mofetil
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
  These patients never switched over to receive mycophenolate mofetil as they were a treatment success at Month 6.
- Methotrexate, Then Mycophenolate Mofetil: first received oral methotrexate
  Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
  then switched over to receive oral mycophenolate mofetil after failing with oral methotrexate
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Followed the same prednisone schedule as described in the Methotrexate only and Mycophenolate Mofetil only groups.
- Mycophenolate Mofetil, Then Methotrexate: first received oral mycophenolate mofetil
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
  then switched over to receive oral mycophenolate mofetil after failing with oral mycophenolate mofetil
  Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Followed the same prednisone schedule as described in the Methotrexate only and Mycophenolate Mofetil only groups.
Period: 0-6 Months
Arm/Group | Methotrexate Only | Mycophenolate Mofetil Only | Methotrexate, Then Mycophenolate Mofetil | Mycophenolate Mofetil, Then Methotrexate
Started | 107 | 109 | 0 | 0
Completed | 96 | 98 | 0 | 0
Not Completed | 11 | 11 | 0 | 0
Period: 6-12 Months
Arm/Group | Methotrexate Only | Mycophenolate Mofetil Only | Methotrexate, Then Mycophenolate Mofetil | Mycophenolate Mofetil, Then Methotrexate
Started | 64 (64 patients were a treatment success on methotrexate at 6 mo and had the option to continue) | 56 (56 patients were a treatment success on mycophenolate mofetil at 6 mo and had the option to continue) | 32 (32 patients failed methotrexate within the first 6 months) | 42 (42 patients failed on mycophenolate mofetil within the first 6 months)
Completed | 60 | 54 | 20 | 29
Not Completed | 4 | 2 | 12 | 13
Not completed — Did not want to switch antimetabolites | 0 | 0 | 9 | 11
Not completed — Adverse Event | 0 | 0 | 3 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in baseline analysis.
Groups:
- Mycophenolate Mofetil: oral mycophenolate mofetil
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [26 to 50] | 41 [31 to 51] | 38 [28 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 60 | 135
  Male | 32 | 49 | 81
Race/Ethnicity, Customized [Number; unit: participants] — Patients could list more than one race.
  participants
    White | 25 | 22 | 47
    Black | 3 | 6 | 9
    Asian | 5 | 6 | 11
    Indian Subcontinent | 70 | 69 | 139
    Native American | 2 | 1 | 3
    Pacific Islander | 1 | 3 | 4
    Middle Eastern | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 4 | 5 | 9
  United States | 22 | 25 | 47
  Mexico | 1 | 2 | 3
  Australia | 11 | 10 | 21
  India | 69 | 67 | 136
Anatomic Location of Uveitis [Count of Participants; unit: Participants]
  Intermediate | 8 | 9 | 17
  Anterior + Intermediate | 15 | 14 | 29
  Posterior | 24 | 25 | 49
  Panuveitis | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Treatment Success at 6 Months (Phase I, 0-6 Months)
Description: Controlled ocular inflammation (≤ 0.5+ anterior chamber cells, ≤ 0.5+ vitreous haze, no active retinal/choroidal lesions in both eyes) with 7.5 mg/day of oral prednisone and ≤ 2 drops/day of topical 1% prednisolone acetate.
Time Frame: 6 Months
Population: All randomized patient with a 6-month visit, or who were declared early treatment failures, are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 96 | 98
Participants | 64 | 56

2. Secondary Outcome: Number of Participants Achieving Treatment Success at 12 Months on Same Medication (Phase I, 6-12 Months)
Description: Controlled ocular inflammation (≤ 0.5+ anterior chamber cells, ≤ 0.5+ vitreous haze, no active retinal/choroidal lesions in both eyes) with 7.5 mg/day of oral prednisone and ≤ 2 drops/day of topical 1% prednisolone acetate in patients who were a treatment success at the primary outcome of 6 months.
Time Frame: 12 Months
Population: Patients who were a treatment success at 6 months and continued in follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Methotrexate: oral methotrexate Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week) Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
Arm/Group | Methotrexate | Mycophenolate Mofetil
Number analyzed (Participants) | 60 | 54
Participants | 48 | 40

3. Secondary Outcome: Number of Participants Achieving Treatment Success After Switching to Other Medication (Phase II, 0-6 Months)
Description: Controlled ocular inflammation (≤ 0.5+ anterior chamber cells, ≤ 0.5+ vitreous haze, no active retinal/choroidal lesions in both eyes) with 7.5 mg/day of oral prednisone and ≤ 2 drops/day of topical 1% prednisolone acetate for patients who crossed over to other medication following treatment failure at 6 months (or earlier).
Time Frame: 6 Months
Population: Patients who switched to the other medication following treatment failure at 6 months (or earlier). Patients were analyzed by the medication that they received in this second phase (Phase II, 0-6 Months).
Measure: Count of Participants; unit: Participants
Groups:
- Switched Over to Methotrexate: oral methotrexate
  Patients were randomized to mycophenolate but were a treatment failure in Phase I, 0-6 Months and switched over to received methotrexate.
  Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
- Switched Over to Mycophenolate Mofetil: oral mycophenolate mofetil
  Patients were randomized to methotrexate but were a treatment failure in Phase I, 0-6 Months and switched over to received mycophenolate mofetil.
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
Arm/Group | Switched Over to Methotrexate | Switched Over to Mycophenolate Mofetil
Number analyzed (Participants) | 29 | 20
Participants | 20 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the primary endpoint (the first 6 months) for each enrolled patient; Phase I, 0-6 Months.
Groups:
- Methotrexate: oral methotrexate
  Patients randomized to receive oral methotrexate in Phase I, 0-6 Months.
  Methotrexate: For the first two weeks, an introductory dose of 15 mg/week (7.5mg BID once a week) orally. After two weeks, the dose will be increased to 25 mg/week (12.5mg BID once a week)
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
- Mycophenolate Mofetil: oral mycophenolate mofetil
  Patients randomized to receive oral mycophenolate mofetil in Phase I, 0-6 Months.
  Mycophenolate mofetil: For the first two weeks, an introductory dose of 500 mg BID orally. After two weeks, the dose will be increased to 1.5 g BID.
  Prednisone: All patients enrolled in the study will be initially taking concomitant oral corticosteroids at 1 mg/kg or 60 mg daily, whichever is less. Initial corticosteroid dose will be continued for 2 to 4 weeks at which point prednisone will be gradually tapered. Prednisone will be tapered to and held at 7.5 mg/day for the first 6 months of the study.
Arm/Group | Methotrexate | Mycophenolate Mofetil
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/109
Serious Adverse Events (participants affected / at risk) | 7/107 | 7/109
Other Adverse Events (participants affected / at risk) | 99/107 | 100/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=107) | Mycophenolate Mofetil (N=109)
Glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
SGOT and SGPT (Blood and lymphatic system disorders) | 3 | 2 — ≥5 times the upper limit of normal of the reference range
Diarrhea (Renal and urinary disorders) | 0 | 1
Disability or permanent damage (Musculoskeletal and connective tissue disorders) | 1 | 0
Hospitalization (General disorders) | 2 | 2
Serious systemic infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Other serious/systemic event (General disorders) | 3 | 1
Death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=107) | Mycophenolate Mofetil (N=109)
Cataract (Eye disorders) | 5 | 2
Suspected/confirmed glaucoma diagnosis (Eye disorders) | 2 | 2
Hypotony (Eye disorders) | 0 | 1 — Intraocular pressure <5 mmHg without structural damage
Ocular hypertension (Eye disorders) | 10 | 13
Peripheral and/or central vitreous hemorrhage (Eye disorders) | 3 | 3
Other ocular event (Eye disorders) | 27 | 26
Creatinine (General disorders) | 1 | 0 — ≥1.5 to <2 mg/dL
Hemoglobin (General disorders) | 2 | 3 — >6.4 to <10 g/dL
Leukocytes (General disorders) | 3 | 1 — >1000 and <2500 µL lasting less than 1 month or absolute neutrophil count (ANC) <1000 but >500
SGOT or SGPT (General disorders) | 14 | 8 — 2 to 5 times the upper limit of normal
Allergic reaction (General disorders) | 14 | 11
Mild congestive heart failure or arrhythmia (Cardiac disorders) | 4 | 2 — Not requiring therapy
Diarrhea (Renal and urinary disorders) | 25 | 24
Dyspnea (General disorders) | 21 | 22
Fatigue (General disorders) | 62 | 59
Fever (General disorders) | 11 | 18 — <103 degrees for 12 hours
Hair loss (General disorders) | 6 | 2
Headache (General disorders) | 55 | 45
Non-serious systemic infection (Infections and infestations) | 25 | 27
Mood changes (Psychiatric disorders) | 33 | 26 — Not requiring therapy
Muscle weakness (Musculoskeletal and connective tissue disorders) | 32 | 26 — No decrease in function
Nausea (General disorders) | 42 | 30
Numbness/tingling (Nervous system disorders) | 25 | 18
Vomiting (General disorders) | 26 | 24
Other systemic (no treatment required) (General disorders) | 65 | 63
Decrease in vision/defective vision (Eye disorders) | 9 | 19
Eye pain (Eye disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT01829295/Prot_SAP_000.pdf